CLINICAL TRIAL: NCT02514213
Title: Phase I, Open-label Trial to Evaluate the Safety and Immunogenicity of INO-5150 Alone or in Combination With INO-9012 in Men With Biochemically Relapsed (PSA) Prostate Cancer
Brief Title: Trial to Evaluate Safety and Immunogenicity of INO-5150 Alone or With INO-9012 in Men With Prostate Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Inovio Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PCa-001
Record Dates: First submitted 2015-07-29; First posted 2015-08-03 (Estimated); Last update posted 2017-12-26 (Actual); Status verified 2017-12

CONDITIONS: Prostate Cancer
Keywords: PSA
MeSH Terms: conditions — Prostatic Neoplasms | interventions — rocakinogene sifuplasmid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Arm A (Experimental): 2mg INO-5150 and electroporation device CELLECTRA®-5P
  Interventions: Biological: 2mg INO-5150 and electroporation device CELLECTRA®-5P; Device: Electroporation using CELLECTRA®-5P
- Arm B (Experimental): 8.5mg INO-5150 and electroporation device CELLECTRA®-5P
  Interventions: Biological: 8.5mg INO-5150 and electroporation device CELLECTRA®-5P; Device: Electroporation using CELLECTRA®-5P
- Arm C (Experimental): 2mg INO-5150 plus 1mg INO-9012 and electroporation device CELLECTRA®-5P
  Interventions: Biological: 2mg INO-5150 plus 1mg INO-9012 and electroporation device CELLECTRA®-5P; Device: Electroporation using CELLECTRA®-5P
- Arm D (Experimental): 8.5mg INO-5150 plus 1mg INO-9012 and electroporation device CELLECTRA®-5P
  Interventions: Biological: 8.5mg INO-5150 plus 1mg INO-9012 and electroporation device CELLECTRA®-5P; Device: Electroporation using CELLECTRA®-5P

INTERVENTIONS:
Biological: 2mg INO-5150 and electroporation device CELLECTRA®-5P — 2mg INO-5150 delivered IM followed by electroporation using CELLECTRA®-5P
  Arms: Arm A
Biological: 8.5mg INO-5150 and electroporation device CELLECTRA®-5P — 8.5 mg INO-5150 delivered IM followed by electroporation using CELLECTRA®-5P
  Arms: Arm B
Biological: 2mg INO-5150 plus 1mg INO-9012 and electroporation device CELLECTRA®-5P — 2mg INO-5150 plus 1 mg INO9012 delivered IM followed by electroporation using CELLECTRA®-5P
  Arms: Arm C
Biological: 8.5mg INO-5150 plus 1mg INO-9012 and electroporation device CELLECTRA®-5P — 8.5mg INO-5150 plus 1 mg INO9012 delivered IM followed by electroporation using CELLECTRA®-5P
  Arms: Arm D
Device: Electroporation using CELLECTRA®-5P — Electroporation device CELLECTRA®-5P

SUMMARY:
This is a phase I, open-label trial to evaluate the safety and immunogenicity of INO 5150 alone or in combination with INO-9012 when delivered intramuscularly (IM) followed by electroporation (EP) in men with biochemically relapsed prostate cancer.

DETAILED DESCRIPTION:
Phase I, open label study of INO-5150 (DNA plasmids encoding prostate specific antigen (PSA) and prostate specific membrane antigen (PSMA)) alone or co-administered with INO-9012 (IL-12 plasmid) delivered intramuscularly followed by EP using the CELLECTRA®-5P device in adult males with biochemically relapsed prostate cancer following definitive local therapy (e.g. prostatectomy, external beam radiation, or brachytherapy). Four injections will be administered to approximately 60 eligible subjects who consent to participate in the study. Subjects will be monitored for safety and immunogenicity through Week 72.

ELIGIBILITY:
Inclusion Criteria:

1. Men aged 18 to 90 years with a histologic diagnosis of prostate cancer;
2. c. Biochemical recurrence following local therapy, either surgery or radiation. Rising PSA defined as:

   * After definitive surgery, e.g.

     * After radical prostatectomy, two PSA measurements of ≥ 1.0 ng/mL at least one week apart;
     * After cryosurgery, two PSA measurements of ≥ 2.0 ng/mL at least one week apart;
     * Other definitive surgical procedures may be permissible upon the approval of the medical monitor OR
   * After radiation therapy (e.g., external beam radiation, brachytherapy, or salvage/adjuvant radiation therapy after surgery), two post radiation PSA measurements level of nadir plus 2.0 ng/mL at least one week apart.;
3. Serum testosterone level:

   i) Subjects with no history of androgen deprivation therapy:
   * A single measurement greater than 150 ng/dL or 5.2 nmol/L within 3 months of enrollment

   ii) Subjects with a history of androgen deprivation therapy (either in adjuvant or biochemical relapse setting):
   * The two most recent measurements of serum testosterone prior to enrollment must fulfill the following criteria:

     * Both measurements are greater than 150 ng/dL or 5.2 nmol/L;
     * The two measurements are spaced at least 14 days apart;
     * Both must be measured within 3 months of enrollment;
4. Normal electro cardio gram (ECG) or ECG with no clinically significant findings;
5. Adequate bone marrow, hepatic, and renal function tests within 30 days prior to enrollment:

   * CBC (except platelets and hemoglobin), serum chemistry, liver panel, and CPK values ≤ Grade 1 abnormality as defined in CTCAE v 4.03 dated June 14, 2010
   * Platelets ≥ 75,000 /mL;
   * Hemoglobin ≥ 9.0 g/dL;
6. No desire or plans to father new children during the study and/or have a prior vasectomy

Exclusion Criteria:

1. PSA doubling time (PSA-DT) of ≤ 3 months, using 2 PSA values at least 4 weeks apart, calculated according to the Memorial Sloan-Kettering Cancer Center nomogram (https://www.mskcc.org/nomograms/prostate/psa-doubling-time);
2. Clinical or radiologic evidence of distant metastatic disease other than small volume (<1.5 cm) nodes, this should be tested within 12 months from enrollment;
3. Receipt of investigational therapy in a clinical trial setting within 30 days of enrollment;
4. Any pre-excitation syndromes, e.g., Wolff-Parkinson-White syndrome;
5. Prior major surgery or radiation therapy within 4 weeks of enrollment;
6. Any prior chemotherapy, except short-course neo-adjuvant or adjuvant chemotherapy that had been stopped for at least 6 weeks prior to Study enrollment;
7. Active AIDS / HIV infection, clinically uncontrolled immune deficiency disorders;
8. Clinically uncontrolled autoimmune disorders, transplant recipients who depend on immunosuppressive therapy, other immunosuppressive conditions including any concurrent condition requiring immunosuppressive/immunomodulating agents;
9. Recipient of any blood product and immunotherapy (such as anti-PD1, anti-PDL-1 and anti-CTLA4) within 3 months of enrollment;

Ages: 18 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2015-07; Primary Completion 2017-12-12 (Actual); Study Completion 2017-12-12 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of INO-5150 alone or with INO-9012 delivered via IM EP ( Incidence of adverse events, Injection site reactions, Changes in safety laboratory parameters) | 72 weeks
  1. Incidence of adverse events (all, severe, [NCI CTCAE v4.03] and serious) classified by system organ class (SOC), preferred term, severity, and relationship to study medication and schedule
  2. Injection site reactions
  3. Changes in safety laboratory parameters .
Antigen specific immune response of INO-5150 alone or with INO-9012 delivered via IM EP | 72 weeks
  Antigen specific cellular immune responses

SECONDARY OUTCOMES:
PSA response rate by PSA testing | 72 weeks
  PSA response

CONTACTS AND LOCATIONS:
Overall Officials: Ildi Csiki, MD, PH.D., Study Director — Inovio Pharmaceuticals
Locations (10):
- United States (10):
  - Chesapeake Urology Research Associates, Baltimore, Maryland
  - Karmanos Cancer Institute, Detroit, Michigan
  - GU Research Network, LLC/ Urology Cancer Center, Omaha, Nebraska
  - Weill Cornell Medical College, New York, New York
  - University of North Carolina Lineberger Cancer Center, Chapel Hill, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Sidney Kimmel Cancer Center - Thomas Jefferson University, Philadelphia, Pennsylvania
  - UPMC, Pittsburgh, Pennsylvania
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - Seattle Cancer Care Alliance, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No
combined results when available will be made available